CLINICAL TRIAL: NCT06582745
Title: Targeted Approach to Langerhans Cell Histiocytosis (LCH) Using MEK Inhibitor, Trametinib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cook Children's Health Care System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-058
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-12

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: LCH; MEK inhibitor; Targeted therapy
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prospective Treatment (Experimental): Trametinib will be administered in 28-day cycles, given once daily or adjusted as per clinical judgment of the treating physician, with a maximum dosage of 2mg daily. Patients will be followed for 4 years after receiving treatment for two years. Patients may continue on the same treatment beyond two years if they and their treating physicians agree to do so in the best interest of the patient.
  Interventions: Drug: Trametinib
- Observation Only (No Intervention): Patients who have been receiving trametinib as a treatment for LCH since January 1, 2020 may be included in an observational chart review to track long-term follow-up.

INTERVENTIONS:
Drug: Trametinib — Participants will be given trametinib as a single agent once a day dosing, with a maximum dose of 2kg. Participants who are able to swallow pills will be given oral tablets. Participants unable to swallow pills will be dispensed the liquid formula concentrate at 0.05mg/mL with dosing of 0.015mg/kg.
  Other Names: Mekinist
  Arms: Prospective Treatment

SUMMARY:
The purpose of this Phase II clinical trial is to establish the safety and effectiveness of trametinib, a targeted therapy, for the treatment of newly or recently diagnosed Langerhans Cell Histiocytosis (LCH) among pediatric patients.

DETAILED DESCRIPTION:
Langerhans cell histiocytosis (LCH) is a rare histiocytic disease derived from the mononuclear phagocytic system, affecting between 2 and 10 cases per one million children under 15 years. Controversy exists as to whether it is a true malignancy or a cancer-like disease, given that the BRAFV600E mutation frequently found in LCH has been found in several cancers as well as in benign nevi. Regardless, among histiocytic disorders, LCH is well-known to result from clonal proliferation of immature cells that can affect a single organ (single system LCH) which may be unifocal or multifocal; or LCH may involve multiple organs which may be limited or widespread. Notably, involvement of specific organs such as the liver, spleen, and bone marrow is typically considered high risk. A biopsy is a critical element for diagnosis as histiocytes with surface expression of CD207 (langerin) and CD1a are a defining characteristic of LCH. In addition to a biopsy of either skin lesion, lymph node, or tumor, standard imaging such as CT, MRI, and PET will be used to assess the extent of disease.

This trial is designed to evaluate treatment of newly diagnosed or relapsed LCH patients with targeted therapy (trametinib). The investigators hypothesize that this will help establish a new treatment for these patients who have historically been treated with cytotoxic chemotherapy that can potentially be associated with serious adverse effects as well as relapse which have typically been noted within two years, therefore justifying the rationale to treat for minimum of two years. This clinical trial will provide an opportunity to assess for adverse events and toxicities associated with trametinib for the treatment of LCH among pediatric patients. Additionally, the investigators will critically analyze the effectiveness of genomic cancer testing through the use of liquid, tumor, and tumor-match next-generation sequencing (NGS) in patients with an LCH diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis/disease status:

  * Patients with newly diagnosed Langerhans cell histiocytosis (LCH) OR
  * Patients with relapsed or refractory disease OR
  * Patients with newly diagnosed or relapsed/refractory disease who are receiving the liquid formula of trametinib OR
  * Patients who have been receiving trametinib as a treatment for LCH since January 1, 2020 may be included in the observational chart review to track long-term follow-up. Eligibility for chart review cohort will include receiving trametinib as treatment.
* Diagnosis confirmed with biopsy prior to start of treatment
* Patient must have adequate cardiac function evident through Echocardiogram (ECHO) and Electrocardiogram (EKG) within 30 days of starting treatment.

  * Shortening fraction of ≥ 27% by echocardiogram or
  * Ejection fraction of ≥ 50% by gated radionuclide study
  * QTC < 480 msec
* Performance status: Patients must have a performance status corresponding to ECOG scores of 0, 1, or 2. Use Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥50% for patients ≤16 years of age.
* Adequate organ and marrow function as defined below:

  * Absolute Neutrophil count ≥ 1,500/μL
  * Platelets ≥ 100x103/μL
  * Total bilirubin ≤ 1.5X ULN for age
  * AST/ALT ≤ 2.5 X ULN for age
  * Serum creatinine based on age/gender
  * Hemoglobin ≥ 8 g/dL

    * Patients with bone marrow disease must have hemoglobin ≥ 8 g/dL with transfusion support allowed
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after the last dose. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Patients diagnosed with Low-Risk True Skin Only or a Single Bone lesion that does not require treatment and will only be observed will not be eligible, with the exception of CNS-risk lesions/special site disease or functionally critical lesions:

  * CNS-risk/special site includes: Sphenoid, Mastoid, Orbital, zygomatic, ethmoid, maxillary, or temporal bones, the cranial fossa, pituitary gland or neurodegenerative disease, odontoid peg, vertebral lesion with intraspinal soft tissue extension
  * Functionally critical: A single lesion not described above which may cause "functionally critical anatomic abnormality" wherein attempts at local therapy would cause unacceptable morbidity. This can be at the discretion of the Principal Investigator.
* Patients whose genetic testing reveals a class 3 MAP2K1 mutation:

  * I103_K104del
  * E102_I103del
  * L98_K104delinsQ
  * L98_I103del
  * I99_K104del
* Patients who present with jaundice at diagnosis.
* Patients who are pregnant or breastfeeding are not eligible. Women of childbearing potential must receive a negative pregnancy test within 14 days of starting treatment or the patient will not be eligible.

  * Patients who are allergic to trametinib
  * Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of patient or parent/legally authorized representative to give written informed consent.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2039-06 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Time to Progression (TTP) | Up to six years
  TTP defined for each participant as the period of time from start of treatment to the manifestation of objective progression, but excluding occurrences of death.
Progression-free Survival (PFS) | Up to six years
  PFS defined for each participant as the time from start of treatment to disease progression (recurrence) or death by any cause in the absence of progression.
Overall Survival (OS) | Up to six years
  OS defined for each participant as the time from the date of first administration until the date of death from any cause. Participants not having an event at the time of analysis will be censored at the date they were last known to be alive.

SECONDARY OUTCOMES:
Response Rate | Up to six years
  The response rate will be defined as the percentage of patients with Complete Response (the disappearance of all signs of LCH in response to treatment), Stable Disease (neither increasing nor decreasing in extent or severity), Partial Response (at least a 30% decrease in the signs of LCH), and Progressive Disease (at least a 20 percent growth in the signs of LCH since the beginning of treatment).
Blood HistioTrak Levels in Participants with BRAF V600E Mutations | Up to six years
  The HistioTrak test is a highly sensitive droplet digital PCR (ddPCR)-based molecular assay designed to measure MRD in patients with BRAF V600E-driven histiocytic and other neoplasms.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Ray, MD, Principal Investigator — Cook Children's Health Care System
Locations (1):
- Cook Children's Health Care System, Fort Worth, Texas, United States

REFERENCES:
- [Background] Stalemark H, Laurencikas E, Karis J, Gavhed D, Fadeel B, Henter JI. Incidence of Langerhans cell histiocytosis in children: a population-based study. Pediatr Blood Cancer. 2008 Jul;51(1):76-81. doi: 10.1002/pbc.21504. PMID 18266220
- [Background] Badalian-Very G, Vergilio JA, Fleming M, Rollins BJ. Pathogenesis of Langerhans cell histiocytosis. Annu Rev Pathol. 2013 Jan 24;8:1-20. doi: 10.1146/annurev-pathol-020712-163959. Epub 2012 Aug 6. PMID 22906202
- [Background] Allen CE, Ladisch S, McClain KL. How I treat Langerhans cell histiocytosis. Blood. 2015 Jul 2;126(1):26-35. doi: 10.1182/blood-2014-12-569301. Epub 2015 Mar 31. PMID 25827831
- [Background] Jouenne F, Chevret S, Bugnet E, Clappier E, Lorillon G, Meignin V, Sadoux A, Cohen S, Haziot A, How-Kit A, Kannengiesser C, Lebbe C, Gossot D, Mourah S, Tazi A. Genetic landscape of adult Langerhans cell histiocytosis with lung involvement. Eur Respir J. 2020 Feb 27;55(2):1901190. doi: 10.1183/13993003.01190-2019. Print 2020 Feb. PMID 31806714
- [Background] Chakraborty R, Hampton OA, Shen X, Simko SJ, Shih A, Abhyankar H, Lim KP, Covington KR, Trevino L, Dewal N, Muzny DM, Doddapaneni H, Hu J, Wang L, Lupo PJ, Hicks MJ, Bonilla DL, Dwyer KC, Berres ML, Poulikakos PI, Merad M, McClain KL, Wheeler DA, Allen CE, Parsons DW. Mutually exclusive recurrent somatic mutations in MAP2K1 and BRAF support a central role for ERK activation in LCH pathogenesis. Blood. 2014 Nov 6;124(19):3007-15. doi: 10.1182/blood-2014-05-577825. Epub 2014 Sep 8. PMID 25202140
- [Background] Vicenzi P, Ray A. Comment on: Langerhans cell histiocytosis with BRAF p.N486_P490del or MAP2K1 p.K57_G61del treated by the MEK inhibitor trametinib. Pediatr Blood Cancer. 2021 Apr;68(4):e28776. doi: 10.1002/pbc.28776. Epub 2020 Oct 21. No abstract available. PMID 33089615
- [Background] Gadner H, Minkov M, Grois N, Potschger U, Thiem E, Arico M, Astigarraga I, Braier J, Donadieu J, Henter JI, Janka-Schaub G, McClain KL, Weitzman S, Windebank K, Ladisch S; Histiocyte Society. Therapy prolongation improves outcome in multisystem Langerhans cell histiocytosis. Blood. 2013 Jun 20;121(25):5006-14. doi: 10.1182/blood-2012-09-455774. Epub 2013 Apr 15. PMID 23589673
- [Background] Morimoto A, Ikushima S, Kinugawa N, Ishii E, Kohdera U, Sako M, Fujimoto J, Bessho F, Horibe K, Tsunematsu Y, Imashuku S; Japan Langerhans Cell Histiocytosis Study Group. Improved outcome in the treatment of pediatric multifocal Langerhans cell histiocytosis: Results from the Japan Langerhans Cell Histiocytosis Study Group-96 protocol study. Cancer. 2006 Aug 1;107(3):613-9. doi: 10.1002/cncr.21985. PMID 16804933
- [Background] Sieni E, Barba C, Mortilla M, Savelli S, Grisotto L, Di Giacomo G, Romano K, Fonda C, Biggeri A, Guerrini R, Arico M. Early Diagnosis and Monitoring of Neurodegenerative Langerhans Cell Histiocytosis. PLoS One. 2015 Jul 15;10(7):e0131635. doi: 10.1371/journal.pone.0131635. eCollection 2015. PMID 26176859
- [Background] Chohan G, Barnett Y, Gibson J, Reddel SW, Barnett MH. Langerhans cell histiocytosis with refractory central nervous system involvement responsive to infliximab. J Neurol Neurosurg Psychiatry. 2012 May;83(5):573-5. doi: 10.1136/jnnp-2011-300575. Epub 2011 Aug 19. No abstract available. PMID 21856693
- [Background] Titgemeyer C, Grois N, Minkov M, Flucher-Wolfram B, Gatterer-Menz I, Gadner H. Pattern and course of single-system disease in Langerhans cell histiocytosis data from the DAL-HX 83- and 90-study. Med Pediatr Oncol. 2001 Aug;37(2):108-14. doi: 10.1002/mpo.1178. PMID 11496348
- [Background] Diamond EL, Durham BH, Ulaner GA, Drill E, Buthorn J, Ki M, Bitner L, Cho H, Young RJ, Francis JH, Rampal R, Lacouture M, Brody LA, Ozkaya N, Dogan A, Rosen N, Iasonos A, Abdel-Wahab O, Hyman DM. Efficacy of MEK inhibition in patients with histiocytic neoplasms. Nature. 2019 Mar;567(7749):521-524. doi: 10.1038/s41586-019-1012-y. Epub 2019 Mar 13. PMID 30867592
- [Background] Haroche J, Cohen-Aubart F, Emile JF, Maksud P, Drier A, Toledano D, Barete S, Charlotte F, Cluzel P, Donadieu J, Benameur N, Grenier PA, Besnard S, Ory JP, Lifermann F, Idbaih A, Granel B, Graffin B, Hervier B, Arnaud L, Amoura Z. Reproducible and sustained efficacy of targeted therapy with vemurafenib in patients with BRAF(V600E)-mutated Erdheim-Chester disease. J Clin Oncol. 2015 Feb 10;33(5):411-8. doi: 10.1200/JCO.2014.57.1950. Epub 2014 Nov 24. PMID 25422482
- [Background] Flaherty KT, Robert C, Hersey P, Nathan P, Garbe C, Milhem M, Demidov LV, Hassel JC, Rutkowski P, Mohr P, Dummer R, Trefzer U, Larkin JM, Utikal J, Dreno B, Nyakas M, Middleton MR, Becker JC, Casey M, Sherman LJ, Wu FS, Ouellet D, Martin AM, Patel K, Schadendorf D; METRIC Study Group. Improved survival with MEK inhibition in BRAF-mutated melanoma. N Engl J Med. 2012 Jul 12;367(2):107-14. doi: 10.1056/NEJMoa1203421. Epub 2012 Jun 4. PMID 22663011
- [Background] Selt F, van Tilburg CM, Bison B, Sievers P, Harting I, Ecker J, Pajtler KW, Sahm F, Bahr A, Simon M, Jones DTW, Well L, Mautner VF, Capper D, Hernaiz Driever P, Gnekow A, Pfister SM, Witt O, Milde T. Response to trametinib treatment in progressive pediatric low-grade glioma patients. J Neurooncol. 2020 Sep;149(3):499-510. doi: 10.1007/s11060-020-03640-3. Epub 2020 Oct 7. PMID 33026636
- [Background] Bouffet E, Hansford JR, Garre ML, Hara J, Plant-Fox A, Aerts I, Locatelli F, van der Lugt J, Papusha L, Sahm F, Tabori U, Cohen KJ, Packer RJ, Witt O, Sandalic L, Bento Pereira da Silva A, Russo M, Hargrave DR. Dabrafenib plus Trametinib in Pediatric Glioma with BRAF V600 Mutations. N Engl J Med. 2023 Sep 21;389(12):1108-1120. doi: 10.1056/NEJMoa2303815. PMID 37733309
- [Background] Eckstein OS, Visser J, Rodriguez-Galindo C, Allen CE; NACHO-LIBRE Study Group. Clinical responses and persistent BRAF V600E+ blood cells in children with LCH treated with MAPK pathway inhibition. Blood. 2019 Apr 11;133(15):1691-1694. doi: 10.1182/blood-2018-10-878363. Epub 2019 Feb 4. No abstract available. PMID 30718231
- [Background] Schwartz LH, Litiere S, de Vries E, Ford R, Gwyther S, Mandrekar S, Shankar L, Bogaerts J, Chen A, Dancey J, Hayes W, Hodi FS, Hoekstra OS, Huang EP, Lin N, Liu Y, Therasse P, Wolchok JD, Seymour L. RECIST 1.1-Update and clarification: From the RECIST committee. Eur J Cancer. 2016 Jul;62:132-7. doi: 10.1016/j.ejca.2016.03.081. Epub 2016 May 14. PMID 27189322
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686